CLINICAL TRIAL: NCT00766012
Title: A Phase I, Single-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics After Multiple Oral Doses of AZD2066 in Japanese Healthy Male Subjects
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics After Multiple Doses of AZD2066 in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Anders Neijber, MD, PhD Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0475C00004
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics; AZD2066; Japanese
MeSH Terms: interventions — AZD2066

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4 dose panels receiving a specified volume of AZD2066 oral solution once daily for 11 days
  Interventions: Drug: AZD2066
- 2 (Placebo Comparator): Included in each dose panel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2066 — Oral solution administered orally once per day on day 1, and then day 3 through to day 12 for the first and second dose panels and day 5 through to day 14 for the third and fourth dose panels. For the fifth and sixth panels, oral solution administered once per day on day 1, and then day 5 through to day 16. Specific dose depends on dose panel.
  Arms: 1
Drug: Placebo — Oral solution administered orally once per day on day 1, and then day 3 through to day 12 for the first and second dose panels and day 5 through to day 14 for the third and fourth dose panels. For the fifth and sixth panels, oral solution administered once per day on day 1, and then day 5 through to day 16.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of AZD2066 when given as multiple doses to Japanese healthy male subjects. Four (4) consecutive multiple-ascending panels are planned. Subjects will start with an initial single dose that is followed by a wash-out period of 48 hours to adequately define the single-dose pharmacokinetics. For the third and forth dose panels, the wash-out period will be extended to be 96 hours to evaluate the safety of subjects. Thereafter the subjects will be dosed once daily for 10 days. Ten (10) subjects will be allocated to each dose panel and randomized to receive either AZD2066 or placebo.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of AZD2066 when given as multiple doses to Japanese healthy male subjects. Four (4) consecutive multiple-ascending panels are planned. Subjects will start with an initial single dose that is followed by a wash-out period of 48 hours to adequately define the single-dose pharmacokinetics. For the third and forth dose panels, the wash-out period will be extended to be 96 hours to evaluate the safety of subjects. Thereafter the subjects will be dosed once daily for 10 days. Furthermore, the study has been expanded to include two additional panels with increment of dose during the multiple dosing period (12 days) in order to obtain sufficient information on safety and tolerability of multiple dosing of AZD2066 in Japanese subjects at higher levels of exposure. Ten (10) subjects will be allocated to each dose panel and randomized to receive either AZD2066 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Healthy Japanese males as judged by the investigator
* Clinically normal physical findings and laboratory values as judged by the investigator and a normal resting ECG.

Exclusion Criteria:

* History of somatic disease/condition, which may interfere with the objectives of the study, as judged by the investigator.
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder.
* Intake of medicine (except occasional paracetamol) within first 2 weeks before first administration of study drug.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2008-09; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability by assessment of vital signs, laboratory variables and ECG | Assessments taken at visit 1 (enrolment), defined time points pre dose and post dose during visit 2 (residential period): days -1 through to day 15 and follow up visit 3

SECONDARY OUTCOMES:
Investigate pharmacokinetic profile (including dose proportionality, degree of accumulation and time dependancy) of AZD2066 in Japanese healthy male subjects | Blood sampling at defined timepoints during residential period and follow-up
Investigate CNS effects of AZD2066 in Japanese healthy male subjects | Psychometric test battery performed at defined timepoints during the residential period. Test on day -1 for training purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Neijber, Study Director — AstraZeneca R&D Södertälje, Sweden; Shin Irie, Principal Investigator — Kyusyu Clinical Phramacology Research Clinic
Locations (1):
- Research SIte, Fukuoka, Japan